CLINICAL TRIAL: NCT04469725
Title: A Phase 2, Open-Label, Multi-Center Study to Evaluate Efficacy, Safety and Tolerability of KN046 in Subjects With Thymic Carcinoma
Brief Title: KN046 (a Humanized PD-L1/CTLA4 Bispecific Single Domain Fc Fusion Protein Antibody) in Subjects With Thymic Carcinoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The termination of this study does not involve safety issues. The overall safety of KN046 is good, and no new safety signals have been found. The decision to terminate this study was made due to the adjustment of the sponsor's development strategy.
Sponsor: Jiangsu Alphamab Biopharmaceuticals Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KN046-205
Record Dates: First submitted 2020-07-07; First posted 2020-07-14 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Thymic Carcinoma
MeSH Terms: conditions — Thymoma

STUDY DESIGN:
Intervention Model Description: subjects enrolled receive KN046
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Thymic carcinoma (Experimental): enrolled subjects will receive KN046 every 2 weeks.
  Interventions: Drug: KN046

INTERVENTIONS:
Drug: KN046 — KN046 5 milligram per kilogram, every 2 weeks

SUMMARY:
This is a Phase 2, open-label, multi-center, single arm study in subjects with advanced thymic carcinoma after failure of platinum-based combination chemotherapy. Subjects should have documented progressive disease while on platinum-based combination chemotherapy. If subjects discontinued platinum-based therapy due to reasons other than progressive disease, subjects should have completed at least 2 cycles of platinum-based combination chemotherapy before the commencement of documented progressive disease. Subjects will be treated with KN046 5 milligram per kilogram every 2 weeks.

ELIGIBILITY:
Inclusion Criteria

* Male or female, ≥18 years
* Pathologically confirmed diagnosis of thymic carcinoma
* Inoperable or metastatic disease
* Had failed at least one regimen containing platinum-based combination chemotherapy for locally advanced unresectable or metastatic disease
* Baseline measurable disease

Exclusion Criteria

* Thymomas, thymolipoma, germ cell tumors, teratomas, seminomas
* Leptomeningeal metastasis or untreated active CNS (central nervous system) metastasis or leptomeningeal metastasis.
* Is currently participating and receiving an investigational drug or has participated in a study of an investigational drug within 4 weeks
* Has received other anti-tumor treatment within 4 weeks
* Major surgery for any reason, except diagnostic biopsy, within 4 weeks of the first administration of trial treatment
* Curative radiation within 3 months of the first dose of trial treatment.
* Subjects receiving immunosuppressive agents (such as steroids) for any reason should be tapered off these drugs before initiation of trial treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2020-12-02 (Actual); Primary Completion 2023-07-07 (Actual); Study Completion 2023-07-07 (Actual)

PRIMARY OUTCOMES:
ORR | up to 2 years
  ORR (best overall response) per RECIST v1.1 calculated as the proportion of subjects with a best overall response defined as confirmed complete response or confirmed partial response (CR+PR) by Independent Review Committee;

SECONDARY OUTCOMES:
DOR | up to 3 years
  DOR (duration of response), calculated as the time from the date of the first documented CR or PR to the first documented progression or death due to underlying cancer;
DCR | up to 3 years
  DCR (disease control rate), calculated as the proportion of subjects with best overall response of CR, PR, or SD (stable disease);
CBR | up to 3 years
  CBR (clinical benefit rate), calculated as the proportion of subjects with best overall response of CR, PR, or SD on at least 24 weeks;
PFS | up to 3 years
  PFS (progression free survival), defined as time from first dose of trial treatment to progression or death due to any cause;
TTR | up to 3 years
  TTR (time to response), calculated as the time from first dose of trial treatment to first documented response (CR+PR);

CONTACTS AND LOCATIONS:
Overall Officials: Xiaolong Fu, MD, Principal Investigator — Shanghai Chest Hospital
Locations (1):
- Shanghai Chest Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Remon J, Girard N, Novello S, de Castro J, Bigay-Game L, Bernabe R, Greillier L, Mosquera J, Cousin S, Juan O, Sampayo M, Besse B. PECATI: A Multicentric, Open-Label, Single-Arm Phase II Study to Evaluate the Efficacy and Safety of Pembrolizumab and Lenvatinib in Pretreated B3-Thymoma and Thymic Carcinoma Patients. Clin Lung Cancer. 2022 May;23(3):e243-e246. doi: 10.1016/j.cllc.2021.07.008. Epub 2021 Jul 20. PMID 34393061